CLINICAL TRIAL: NCT07088419
Title: Tinidazole for Mycoplasma Genitalium-Urethritis in the Public Health - Seattle & King County Sexual Health Clinic
Brief Title: "Sexual Health Assessment of TinidaZole Against M. Genitalium (SHAZAM)"
Acronym: SHAZAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Principal Investigator, Lisa Manhart, Professor, Epidemiology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021780; None, N/A (Other: Hologic, Inc)
Record Dates: First submitted 2025-05-28; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mycoplasma Genitalium; Non-gonococcal Urethritis (NGU)
Keywords: Sexually Transmitted Disease (STD); Sexually Transmitted Infection (STI); Mycoplasma genitalium; Tinidazole; Non-gonococcal urethritis (NGU)
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Tinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tinidazole (Experimental): Single Arm
  Interventions: Drug: Tinidazole

INTERVENTIONS:
Drug: Tinidazole — 2 grams orally on day one followed by 500mg orally twice daily on days 2-10

SUMMARY:
The objective is to estimate the efficacy of tinidazole for the treatment of Mycoplasma genitalium (MG) among male patients who have been diagnosed with non-gonococcal urethritis (NGU) at the Public Health - Seattle &King County (PHSKC) Sexual Health Clinic (SHC). Tinidazole was approved by the Food and Drug Administration (FDA) in May 2004 to treat other infections (i.e., trichomoniasis, giardiasis, amebiasis, bacterial vaginosis) but has not been systematically tested for effectiveness against M. genitalium. The dosing that the investigators are proposing does not significantly increase the risk associated with taking tinidazole and this investigation meets criteria for an IND exemption.

DETAILED DESCRIPTION:
To estimate the efficacy of tinidazole for treating M. genitalium among people male sex at birth (men) diagnosed with NGU, the investigators will enroll men with NGU attending an urban sexual health clinic who have a positive test for M. genitalium. Prior to enrollment, men with NGU will have received syndromic therapy for NGU consisting of doxycycline 100mg orally twice daily for 7 days. After enrollment men with NGU will receive tinidazole 2 grams orally on day one followed by 500mg orally twice daily on days 2-10. Participants will undergo a test of cure 21 days after completing the tinidazole regimen to determine whether M. genitalium has been eradicated (microbiologic cure). Remnant urine specimens from the NGU diagnosis visit will be used to perform culture and minimum inhibitory concentration (MIC) assessment, and will undergo quantitative PCR (qPCR) to determine initial organism load. Urine specimens collected at the initiation of tinidazole therapy and at the test of cure will also undergo culture, MIC assessment, and qPCR .

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Clinical diagnosis of NGU
* Urogenital MG documented by a positive NAAT in the prior 7 days
* Fluent in English
* Assigned male at birth
* Attending the PHSKC SHC
* Able to provide informed consent
* Able to undergo a test of cure (TOC) 21 days after completing the tinidazole regimen

Exclusion Criteria:

* Known allergy to tinidazole
* Other contraindications to tinidazole
* At the clinician's discretion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Microbiologic cure of M. genitalium | Day 38
  Microbiologic cure of M. genitalium will be determined at a test of cure visit. Microbiologic cure will be defined as a negative test for M. genitalium in a urine specimen using a nucleic acid amplification test.

SECONDARY OUTCOMES:
Antimicrobial susceptibility to tinidazole (MIC levels) | baseline; day 7; day 38
  The investigators will culture M. genitalium and determine the MIC range for tinidazole.
Antimicrobial susceptibility to tinidazole (resistance associated mutations) | baseline; day 7; day 38
  The investigators will use selective whole genome amplification to identify potential tinidazole resistance associated mutations (TRAMs).
Association of high MIC levels with treatment failure | Day 38
  Using results from Secondary Outcome Measure #2 (culture of M. genitalium from determination of the minimum inhibitory concentration for tinidazole), the investigators will perform statistical analyses to determine if MIC levels are correlated with treatment failure.
Association of tinidazole resistance-associated mutations with treatment failure | Day 38
  Using results from Secondary Outcome Measure #3, the investigators will use statistical methods to determine if specific tindazole resistance-associated mutatons are correlated with microbiologic cure.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Manhart, PhD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Public Health - Seattle & King County Sexual Health Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will adhere to sponsor reporting requirements for IPD. The investigators will share anonymized data to qualified investigators who request it upon IRB approval. The investigators will have the University of Washington IRB review other requests for sharing IPD.